CLINICAL TRIAL: NCT06801743
Title: WHEN DO WE HAVE to PERFORM CARDIAC MAGNETIC RESONANCE in PATIENTS REFERRED for PREMATURE VENTRICULAR COMPLEXES by THEIR CARDIOLOGISTS
Acronym: IRMESV
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0169
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Premature Ventricular Complexes; Ventricular Arythmias; Cardiac Magnetic Resonance Imaging; Focal or Diffuse Fibrosis; Structural Heart Disease; Idiopathic
Keywords: premature ventricular complexes; ventricular arythmias; cardiac magnetic resonance; focal or diffuse fibrosis; structural heart disease; idiopathic
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Premature ventricular complexes (PVC) are a common entity affecting approximatively 20% of the general population. It can be discovered incidentally on electrocardiogram (ECG) or associated with symptoms with a wide spectrum from palpitations, chest pain, to syncope.

The initial and non invasive assessment includes holter ECG monitoring, a transthoracic echocardiography (TTE) and an exercise stress test to rule out structural heart disease (SHD), and referred to as benign or "idiopathic" ventricular arrhythmias (IVA).

However, these exams may fail to identify subtle myocardial abnormalities such as arrhythmogenic right ventricle dysplasia (ARVD), apical hypertrophic cardiomyopathy, healed myocarditis, ischemic or non-ischemic cardiomyopathies.

Cardiac magnetic resonance (CMR) imaging is the gold standard modality to assess regional and global ventricular function. It is also a unique modality to non-invasively detect myocardial edema, myocardial fatty replacement, focal and diffuse fibrosis and could potentially identify SHD in patients with PVC.

However, the role of CMR is uncertain, recommended in case of atypical presentation or when the initial assessment can't exclude a cardiomyopathy (recommendations class IIa).

This study sought to determine whether and when CMR can be performed to provide diagnosis or prognostic information complementary to initial assessment in patients referred for PVC by their cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* patients with PVC who have performed ECG, Holter ECG and a CMR

Exclusion Criteria:

* patient showing opposition tu use his personal data for the reseach,
* patient unable to express his opposition,
* patient deprived of liberty,
* patient with language issues (speaking or writing French)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with PVC who have performed ECG, Holter ECG and a CMR
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of myocardial abnormalities identified by CMR | 1 day
  Composite endpoint of myocardial abnormalities identified by CMR including dilated cardiomyopathy, hypertrophic cardiomyopathy, ischemic cardiomyopathy, ventricular non-compaction, ARVD, myocarditis, pericarditis, sarcoidosis, amyloidosis, Fabry disease

SECONDARY OUTCOMES:
number of criteria to predict myocardial abnormalities on CMR | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospital-Universitaire d'Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No